CLINICAL TRIAL: NCT04199338
Title: The Effect of Web Based Education Based on Self-Care Deficiency Theory on Self-Care Power and Self-Efficacy and Perceived Social Support in Adults Patients Receiving Peritoneal Dialysis Treatment
Brief Title: The Effect of Web Based Education Based on Self-Care Deficiency Theory on Self-Care Power and Self-Efficacy and Perceived Social Support in Patients Receiving Peritoneal Dialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hatice CEYLAN, Principal Investigator, Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: University of Akdeniz
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Self-Care; Self Efficacy; Perceived Social Support; Peritoneal Dialysis
Keywords: peritoneal dialysis,; Orem' self defiency theory; Nursing; Randomized Controlled Trial; Renal Dialysis

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled study
Masking Description: Only participant masking was performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Randomized (Experimental): Randomized
  Interventions: Other: The Effect of Web Based Education Based on Self-Care Deficiency Theory on Self-Care Power and Self-Efficacy and Perceived Social Support in Patients Receiving Peritoneal Dialysis

INTERVENTIONS:
Other: The Effect of Web Based Education Based on Self-Care Deficiency Theory on Self-Care Power and Self-Efficacy and Perceived Social Support in Patients Receiving Peritoneal Dialysis — In the study, which will last for 3 months, the patients in the intervention group will receive pre-test Web-based training based on the Self-Care Deficiency Theory. And an intervention group will be expected to use the website weekly. Also weekly reminder messages will be sent regularly.
  Following the final test, individuals in the enterprise group will be asked to evaluate their views on the website in writing with the WAMMI test.
  Other Names: Web Based Education Based on Self-Care Deficiency Theory

SUMMARY:
Web-based training based on the Self-Care Deficiency Theory has an effect on increasing self-care in in patients undergoing peritoneal dialysis.

Web-based training based on Self-Care Deficiency Theory has an effect on increasing self-efficacy in patients undergoing peritoneal dialysis.

Web-based education based on Self-Care Deficiency Theory has an effect on increasing perceived social support level in patients undergoing peritoneal dialysis.

DETAILED DESCRIPTION:
In the study, which will last for 3 months, the patients in the intervention group will receive pre-test Web-based training based on the Self-Care Deficiency Theory. And an intervention group will be expected to use the website weekly. Also weekly reminder messages will be sent regularly.

Following the final test, individuals in the enterprise group will be asked to evaluate their views on the website in writing with the WAMMI test.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were receive peritoneal dialysis at Akdeniz University Hospital.
* Patients who receiving peritoneal dialysis treatment for at least one months
* Patients who were over 18 years of age,
* Patients who had orientation of individual, place and time
* Patients who were literate
* Patients who has Internet at home
* Patients who has computer or mobile phone
* Patients who no barriers to written or verbal communication
* Patients who agree to participate in the study

Exclusion Criteria:

* Diagnosis of psychiatric illness
* Malignancy diagnosed
* Visually and hearing impaired

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Has an effect on self-care power. | 3 months
  Self-care Power Scale is a Likert-type scale that consists of 25 items and is scored from 0-2.
  In the evaluation, low scores are considered to be good, high scores are not good self-care power.The scale was developed in Turkey.
Has an effect on self-efficacy. | 3 months
  Self-efficacy scale have 10 expressions in the Turkish form and each receives scores ranging from 1 to 4. The lowest score obtained from the scale is evaluated as 10 and the highest score as 40. Self-efficacy score increases as the scale score increases.The scale was developed in Turkey.
Has an effect on perceived social support | 3 months
  The perceived social support scale consisted of 12 items and each consisted of 3 groups regarding the source of the support consisting of 4 items. The higher the score, the higher the perceived social support.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep ÖZER, PhD, RN, Study Director — Akdeniz University
Locations (1):
- Hatice CEYLAN, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will share
Supporting Information: Study Protocol, SAP
Time Frame: starting 1 months after publication
Access Criteria: all people access.

REFERENCES:
- [Background] Rambod M, Rafii F. Perceived social support and quality of life in Iranian hemodialysis patients. J Nurs Scholarsh. 2010 Sep 1;42(3):242-9. doi: 10.1111/j.1547-5069.2010.01353.x. PMID 20738734
- [Background] Plantinga LC, Fink NE, Harrington-Levey R, Finkelstein FO, Hebah N, Powe NR, Jaar BG. Association of social support with outcomes in incident dialysis patients. Clin J Am Soc Nephrol. 2010 Aug;5(8):1480-8. doi: 10.2215/CJN.01240210. Epub 2010 Apr 29. PMID 20430940
- [Background] O'Shaughnessy M. Application of Dorothea Orem's Theory of Self-Care to the Elderly Patient on Peritoneal Dialysis. Nephrol Nurs J. 2014 Sep-Oct;41(5):495-7. PMID 26295092
- [Background] Ramezani T, Sharifirad G, Rajati F, Rajati M, Mohebi S. Effect of educational intervention on promoting self-care in hemodialysis patients: Applying the self-efficacy theory. J Educ Health Promot. 2019 Mar 14;8:65. doi: 10.4103/jehp.jehp_148_18. eCollection 2019. PMID 31008132